CLINICAL TRIAL: NCT05394350
Title: A Phase 1/Phase 2 Study to Evaluate the Safety and Tolerability of MK-1088 as Monotherapy and in Combination With Pembrolizumab in Participants With Advanced Solid Tumors
Brief Title: A Study of MK-1088 as Monotherapy and in Combination With Pembrolizumab in Participants With Advanced Solid Tumors (MK-1088-002)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1088-002; MK-1088-002 (Other: Merck); 2022-502288-40-00 (Registry Identifier: CTIS (EU)); 2021-006712-93 (EudraCT Number)
Record Dates: First submitted 2022-05-23; First posted 2022-05-27 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- MK-1088 100 mg (Experimental): Participants received MK-1088 daily (QD) orally at 100 mg on days 1-21 of each 21-day cycle for up to 35 cycles (up to ~24 months).
  Interventions: Drug: MK-1088
- MK-1088 200 mg (Experimental): Participants received MK-1088 (QD) orally at 200 mg on days 1-21 of each 21-day cycle for up to 35 cycles (up to ~24 months)
  Interventions: Drug: MK-1088
- MK-1088 400 mg (Experimental): Participants received MK-1088 (QD) orally at 400 mg on days 1-21 of each 21-day cycle for up to 35 cycles (up to ~24 months)
  Interventions: Drug: MK-1088
- MK-1088 600 mg (Experimental): Participants received MK-1088 (QD) orally at 600 mg on days 1-21 of each 21-day cycle for up to 35 cycles (up to ~24 months)
  Interventions: Drug: MK-1088
- MK-1088 100 mg + Pembrolizumab (Experimental): Participants received MK-1088 daily (QD) orally at 100 mg on days 1-21 of each 21-day cycle plus pembrolizumab at 200 mg intravenous (IV) infusion every 3 weeks (Q3W), on Day 1 of each 21-day cycle for up to 35 cycles (up to ~24 months)
  Interventions: Drug: MK-1088; Biological: Pembrolizumab
- MK-1088 200 mg + Pembrolizumab (Experimental): Participants received MK-1088 daily (QD) orally at 200 mg on days 1-21 of each 21-day cycle plus pembrolizumab at 200 mg intravenous (IV) infusion every 3 weeks (Q3W), on Day 1 of each 21-day cycle for up to 35 cycles (up to ~24 months)
  Interventions: Drug: MK-1088; Biological: Pembrolizumab

INTERVENTIONS:
Drug: MK-1088 — Oral Tablet
Biological: Pembrolizumab — IV Infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: MK-1088 100 mg + Pembrolizumab; MK-1088 200 mg + Pembrolizumab

SUMMARY:
The study will evaluate the safety, tolerability, and pharmacokinetics (PK) of MK-1088 in monotherapy and in combination with pembrolizumab in participants with advanced solid tumors who have not responded to conventional therapy. The effect of MK-1088 on tumor size will also be examined.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Has a histologically- or cytologically-confirmed diagnosis of advanced/metastatic solid tumor by pathology report and have received, have been intolerant to, or have been ineligible for treatment known to confer clinical benefit
* For metastatic castrate-resistant prostate cancer (mCRPC) only: (1) Must have previously received docetaxel, prior treatment with one other chemotherapy is allowed as well as up to 2 second-generation hormonal manipulations and (2) have prostate cancer progression within 6 months before screening, as determined by the investigator
* If human immunodeficiency virus (HIV) positive, has well-controlled HIV on anti-retroviral therapy (ART)

Exclusion Criteria:

* Has had chemotherapy, definitive radiation, or biological cancer therapy within 4 weeks (2 weeks for palliative radiation) before the first dose of study intervention
* Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years
* Has clinically active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has an active infection requiring therapy
* Has a history of interstitial lung disease
* Has a history of (noninfectious) pneumonitis that required steroids or current pneumonitis
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* Has concurrent active Hepatitis B and Hepatitis C virus infection
* Has HIV with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has not fully recovered from any effects of major surgery without significant detectable infection
* Has a history or current evidence of a gastrointestinal (GI) condition or impaired liver function or diseases that in the opinion of the investigator may significantly alter the absorption or metabolism of oral medications
* Has clinically significant cardiovascular disease within 12 months from first dose of study intervention, including New York Health Association (NYHA) Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability
* Has a corrected QT interval using Fridericia's Correction Formula (QTcF) >470 msec
* Has history of an allogeneic stem cell transplant or a solid organ transplant.
* Has received prior systemic anticancer therapy including investigational agents within 4 weeks before allocation
* Has received prior radiotherapy within 2 weeks of start of study intervention, or had radiation-related toxicities requiring corticosteroids
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Has a "superscan" bone scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (13):
- United States (3):
  - University of Miami Hospital and Clinics, Sylvester Cancer Center ( Site 0103), Miami, Florida
  - Laura and Isaac Perlmutter Cancer Center ( Site 0102), New York, New York
  - South Texas Accelerated Research Therapeutics (START) ( Site 0101), San Antonio, Texas
- Canada (2):
  - Princess Margaret Cancer Centre-Division of Medical Oncology and Hematology ( Site 0201), Toronto, Ontario
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus ( Site 0, Québec, Quebec
- Denmark (3):
  - Rigshospitalet ( Site 0500), Copenhagen, Capital Region
  - Herlev and Gentofte Hospital ( Site 0501), Copenhagen, Capital Region
  - Odense Universitetshospital ( Site 0502), Odense, Region Syddanmark
- Israel (2):
  - Rambam Health Care Campus-Oncology Division ( Site 0300), Haifa
  - Hadassah Medical Center ( Site 0302), Jerusalem
- Switzerland (3):
  - Cantonal Hospital St.Gallen ( Site 0403), Sankt Gallen, Canton of St. Gallen
  - Ospedale Regionale Bellinzona e Valli ( Site 0400), Bellinzona, Canton Ticino
  - Kantonsspital Graubünden-Medizin ( Site 0402), Chur, Kanton Graubünden

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26166&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was closed to enrollment on 04-MAY-2023 for all participants, and no participants remain on treatment with MK-1088. Part 2 of the study was not initiated.
Pre-assignment Details: Per protocol two participants who progressed by radiographic evaluation on monotherapy with MK-1088 at the investigator's discretion and after consultation with the Sponsor, switched over to combination treatment arm of MK-1088 and pembrolizumab.
Period: Overall Study
Arm/Group | MK-1088 100 mg | MK-1088 200 mg | MK-1088 400 mg | MK-1088 600 mg | MK-1088 100 mg + Pembrolizumab | MK-1088 200 mg + Pembrolizumab
Started | 3 | 3 | 11 | 3 | 3 | 4
Switch Over to MK-1088 100 mg + Pembrolizumab | 0 | 1 | 1 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 11 | 3 | 3 | 4
Not completed — Death | 2 | 2 | 4 | 0 | 1 | 0
Not completed — Study terminated by sponsor | 1 | 1 | 7 | 3 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-1088 100 mg | MK-1088 200 mg | MK-1088 400 mg | MK-1088 600 mg | MK-1088 100 mg + Pembrolizumab | MK-1088 200 mg + Pembrolizumab | Total
Number analyzed (Participants) | 3 | 3 | 11 | 3 | 3 | 4 | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.7 (13.6) | 58.7 (24.8) | 59.5 (13.5) | 62.7 (4.9) | 61.0 (10.1) | 55.8 (11.6) | 60.1 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 5 | 2 | 1 | 1 | 10
  Male | 2 | 3 | 6 | 1 | 2 | 3 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 0 | 1 | 3
  Not Hispanic or Latino | 2 | 3 | 10 | 3 | 3 | 3 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 3 | 3 | 11 | 2 | 1 | 4 | 24
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing a Dose-limiting Toxicity (DLT)
Description: A DLT is defined as an event with toxicity including the type, severity, time of onset, time of resolution, and the probable association with study treatment that are not due to pre-existing conditions as defined by the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE 5.0). Per protocol participants who switched over from MK-1088 monotherapy into MK-1088 100 mg + Pembrolizumab combination therapy completed the DLT evaluation period in the monotherapy arm assigned. Percentage of participants who experienced a DLT are presented.
Time Frame: Up to 21 days
Population: All participants who received at least one dose of study intervention and met the criteria for DLT evaluability
Measure: Number; unit: Percentage of Participants
Groups:
- MK-1088 100 mg + Pembrolizumab Switchover: Participants who progressed by radiographic evaluation on monotherapy with MK-1088 and switched over to combination therapy received MK-1088 daily (QD) orally at 100 mg on days 1-21 of each 21-day cycle plus pembrolizumab at 200 mg intravenous (IV) infusion every 3 weeks (Q3W), on Day 1 of each 21-day cycle for up to 35 cycles (up to ~24 months)
Arm/Group | MK-1088 100 mg | MK-1088 200 mg | MK-1088 400 mg | MK-1088 600 mg | MK-1088 100 mg + Pembrolizumab | MK-1088 200 mg + Pembrolizumab | MK-1088 100 mg + Pembrolizumab Switchover
Number analyzed (Participants) | 3 | 3 | 11 | 3 | 3 | 4 | 0
Percentage of Participants | 0.0 | 0.0 | 9.09 | 0.0 | 0.0 | 0.0 |

2. Primary Outcome: Percentage of Participants Experiencing an Adverse Event (AE)
Description: An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. Safety data from participants who experienced disease progression in the monotherapy arm and crossed over into the combination arm are summarized in their initial monotherapy dose group until the time of cross over and are summarized separately thereafter. The percentage of participants who experienced an AE are presented.
Time Frame: Up to ~13 months
Population: All participants who received at least one dose of study intervention
Measure: Number; unit: Percentage of participants
Arm/Group | MK-1088 100 mg | MK-1088 200 mg | MK-1088 400 mg | MK-1088 600 mg | MK-1088 100 mg + Pembrolizumab | MK-1088 200 mg + Pembrolizumab | MK-1088 100 mg + Pembrolizumab Switchover
Number analyzed (Participants) | 3 | 3 | 11 | 3 | 3 | 4 | 2
Percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

3. Primary Outcome: Percentage of Participants Discontinuing Study Treatment Due to an AE
Description: An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. Safety data from participants who experienced disease progression in the monotherapy arm and crossed over into the combination arm are summarized in their initial monotherapy dose group until the time of cross over and are summarized separately thereafter. The percentage of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to ~10 months
Population: All participants who received at least one dose of study intervention
Measure: Number; unit: Percentage of participants
Arm/Group | MK-1088 100 mg | MK-1088 200 mg | MK-1088 400 mg | MK-1088 600 mg | MK-1088 100 mg + Pembrolizumab | MK-1088 200 mg + Pembrolizumab | MK-1088 100 mg + Pembrolizumab Switchover
Number analyzed (Participants) | 3 | 3 | 11 | 3 | 3 | 4 | 2
Percentage of participants | 0.0 | 0.0 | 9.1 | 0.0 | 66.7 | 75.0 | 0.0

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUC) of MK-1088
Description: AUC of MK-1088 determined by blood samples collected pre-dose and at designated timepoints post-dose are presented.
Time Frame: Pre-dose and 1, 2, 4, and 8 hours post-dose on Cycle 1 Day 1 and Cycle 2 Day 1; Pre-dose on Cycle 1 Day 2 and Cycle 2 Day 2; Pre-dose on Cycle 3, Cycle 4 and every 4 cycles up to ~3.5 months. Each cycle = 21 days
Population: All participants who complied with the protocol sufficiently to ensure that their data will be likely to show the effects of treatment, according to the underlying scientific model. Only the per protocol analysis set (excluding the data from the participants after switching over to MK-1088 100 mg and Pembrolizumab) were analyzed for pharmacokinetic (PK) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μmol/L
Arm/Group | MK-1088 100 mg | MK-1088 200 mg | MK-1088 400 mg | MK-1088 600 mg | MK-1088 100 mg + Pembrolizumab | MK-1088 200 mg + Pembrolizumab | MK-1088 100 mg + Pembrolizumab Switchover
Number analyzed (Participants) | 3 | 3 | 11 | 3 | 3 | 4 | 0
hr*μmol/L
  Cycle 1 | 31.9 (105.2) | 26.1 (95.1) | 98.4 (38.5) | 99.4 (43.9) | 21.8 (51.2) | 49.3 (50.8) |
  Cycle 2: number analyzed (Participants) | 2 | 3 | 5 | 3 | 3 | 3 | 0
  Cycle 2 | 39.0 (46.6) | 39.5 (145.4) | 197.0 (46.4) | 188.0 (90.6) | 29.7 (97.1) | 102.0 (17.6) |

5. Secondary Outcome: Maximum Plasma Concentration (Cmax) of MK-1088
Description: Cmax of MK-1088 determined by blood samples collected pre-dose and at designated timepoints post-dose are presented.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μmol/L
Arm/Group | MK-1088 100 mg | MK-1088 200 mg | MK-1088 400 mg | MK-1088 600 mg | MK-1088 100 mg + Pembrolizumab | MK-1088 200 mg + Pembrolizumab | MK-1088 100 mg + Pembrolizumab Switchover
Number analyzed (Participants) | 3 | 3 | 11 | 3 | 3 | 4 | 0
μmol/L
  Cycle 1 | 2.58 (61.8) | 2.17 (50.8) | 6.63 (36.7) | 7.70 (46.4) | 1.41 (62.4) | 3.29 (83.1) |
  Cycle 2: number analyzed (Participants) | 2 | 3 | 5 | 3 | 3 | 3 | 0
  Cycle 2 | 2.82 (31.9) | 3.27 (92.0) | 11.6 (31.8) | 11.6 (79.9) | 1.80 (117.4) | 6.32 (30.2) |

6. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) or Prostate Cancer Working Group (PCWG)-Modified RECIST 1.1 as Assessed by Investigator
Description: ORR is defined as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 or Prostate Cancer Working Group (PCWG)-modified RECIST 1.1 as assessed by investigator. Efficacy data from participants who experienced disease progression in the monotherapy arm and crossed over into the combination arm will be summarized in their initial monotherapy dose group until the time of cross over and will be summarized separately thereafter. The percentage of participants who experience a CR or PR as assessed by the investigator based on RECIST 1.1 is presented.
Time Frame: Up to ~13 months
Population: All participants with a screening/baseline scan that showed measurable disease by the investigator's assessment, and received at least 1 dose of study intervention
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MK-1088 100 mg | MK-1088 200 mg | MK-1088 400 mg | MK-1088 600 mg | MK-1088 100 mg + Pembrolizumab | MK-1088 200 mg + Pembrolizumab | MK-1088 100 mg + Pembrolizumab Switchover
Number analyzed (Participants) | 2 | 3 | 11 | 3 | 3 | 4 | 2
Percentage of participants | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 84.2]

ADVERSE EVENTS:
Time Frame: Death and adverse events up to ~13 months
Description: Every participant is counted a single time for each applicable serious adverse event. MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to the drug are excluded.
Groups:
- MK 1088 100 mg + Pembrolizumab: Participants received MK-1088 daily (QD) orally at 100 mg on days 1-21 of each 21-day cycle plus pembrolizumab at 200 mg intravenous (IV) infusion every 3 weeks (Q3W), on Day 1 of each 21-day cycle for up to 35 cycles (up to ~24 months)
- MK-1088 100 mg + Pembrolizumab Swicthover: Participants who progressed by radiographic evaluation on monotherapy with MK-1088 and switched over to combination therapy received MK-1088 daily (QD) orally at 100 mg on days 1-21 of each 21-day cycle plus pembrolizumab at 200 mg intravenous (IV) infusion every 3 weeks (Q3W), on Day 1 of each 21-day cycle for up to 35 cycles (up to ~24 months)
Arm/Group | MK-1088 100 mg | MK-1088 200 mg | MK-1088 400 mg | MK-1088 600 mg | MK 1088 100 mg + Pembrolizumab | MK-1088 200 mg + Pembrolizumab | MK-1088 100 mg + Pembrolizumab Swicthover
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/3 | 4/11 | 0/3 | 1/3 | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 6/11 | 1/3 | 2/3 | 2/4 | 0/2
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 11/11 | 3/3 | 3/3 | 4/4 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1088 100 mg (N=3) | MK-1088 200 mg (N=3) | MK-1088 400 mg (N=11) | MK-1088 600 mg (N=3) | MK 1088 100 mg + Pembrolizumab (N=3) | MK-1088 200 mg + Pembrolizumab (N=4) | MK-1088 100 mg + Pembrolizumab Swicthover (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1088 100 mg (N=3) | MK-1088 200 mg (N=3) | MK-1088 400 mg (N=11) | MK-1088 600 mg (N=3) | MK 1088 100 mg + Pembrolizumab (N=3) | MK-1088 200 mg + Pembrolizumab (N=4) | MK-1088 100 mg + Pembrolizumab Swicthover (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 4 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (4) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The decision to close study enrollment was based on review of data from the dose escalation phase and Sponsor prioritization. The decision to stop enrollment was not due to any safety concerns, and there were no safety signals observed during the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/50/NCT05394350/Prot_SAP_000.pdf